CLINICAL TRIAL: NCT01059682
Title: A Multi-Center, Double-blind, Randomized, Placebo Controlled, Parallel Group Study of the Effect of Dalcetrapib on Atherosclerotic Disease Progression As Measured by Coronary Intravascular Ultrasound, Carotid B-Mode Ultrasound and Coronary Angiography
Brief Title: A Study of the Effect of Dalcetrapib on Artherosclerotic Disease in Patients With Coronary Artery Disease
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Termination of the clinical development program by the Sponsor
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NC22703
Record Dates: First submitted 2010-01-29; First posted 2010-02-01 (Estimated); Results first posted 2020-03-24 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases | interventions — dalcetrapib

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Dalcetrapib (Experimental)
  Interventions: Drug: Dalcetrapib
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dalcetrapib — Dalcetrapib 600 mg orally once daily
  Arms: Dalcetrapib
Drug: Placebo — Placebo orally once daily
  Arms: Placebo

SUMMARY:
This multicenter, double-blind, randomized, placebo-controlled study will evaluate the effect of dalcetrapib 600 mg on artherosclerotic disease progression, lipid profile and biomarker profile and long-term safety profile of dalcetrapib in patients with coronary artery disease. Atherosclerotic disease progression will be measured 1. Coronary Intravascular Ultrasound (IVUS), Quantitative Coronary Angiography 2. Carotid B-Mode Ultrasound Intima Medial Thickness (IMT) and total plaque volume in subjects undergoing coronary angiography who have coronary artery disease (CAD). Patients will be randomized to receive dalcetrapib 600 mg orally once a day or placebo. The anticipated time on study treatment will be 24 months. The target sample size is 800-1000 patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients over the age of 18 years
* Angiographic evidence of coronary artery disease
* Ultrasound evidence of carotid artery disease
* Treated appropriately for dyslipidemia

Exclusion Criteria:

* Previous exposure to any cholesteryl ester transfer protein (CETP) inhibitor or CETP-vaccine within the last 3 months before study start
* Previous coronary artery bypass graft surgery (CABG) or probable need for CABG in the next 24 months
* Myocardial infarction in the target coronary artery for IVUS between the initial IVUS examination and randomization
* Patients who have symptomatic congestive heart failure at baseline (New York Heart Association class III or IV)
* Severe anemia
* Uncontrolled hypertension
* Poorly controlled diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 936 (Actual)
Dates: Start 2010-01; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (95):
- United States (39):
  - Los Angeles, California
  - Torrance, California
  - Boulder, Colorado
  - Greeley, Colorado
  - Littleton, Colorado
  - Hartford, Connecticut
  - Atlantis, Florida
  - Fort Lauderdale, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - Sarasota, Florida
  - Tampa, Florida
  - Decatur, Georgia
  - Chicago, Illinois
  - Elkhart, Indiana
  - Louisville, Kentucky
  - Columbia, Maryland
  - Salisbury, Maryland
  - Boston, Massachusetts
  - Ann Arbor, Michigan
  - Kalamazoo, Michigan
  - Midland, Michigan
  - Muskegon, Michigan
  - Petoskey, Michigan
  - Duluth, Minnesota
  - Rochester, Minnesota
  - Kansas City, Missouri
  - Paramus, New Jersey
  - New York, New York
  - Rochester, New York
  - Chapel Hill, North Carolina
  - Toledo, Ohio
  - Hershey, Pennsylvania
  - Providence, Rhode Island
  - Germantown, Tennessee
  - Oak Ridge, Tennessee
  - Dallas, Texas
  - Houston, Texas
  - Richmond, Virginia
- Canada (36):
  - Calgary, Alberta
  - Edmonton, Alberta
  - New Westminster, British Columbia
  - Vancouver, British Columbia
  - Victoria, British Columbia
  - Saint John, New Brunswick
  - St. John's, Newfoundland and Labrador
  - Halifax, Nova Scotia
  - Brampton, Ontario
  - Burlington, Ontario
  - Cambridge, Ontario
  - Hamilton, Ontario
  - Kitchener, Ontario
  - London, Ontario
  - Mississauga, Ontario
  - Newmarket, Ontario
  - Oshawa, Ontario
  - Ottawa, Ontario
  - Scarborough Village, Ontario
  - Toronto, Ontario
  - Chicoutimi, Quebec
  - Fleurimont, Quebec
  - Gatineau, Quebec
  - Greenfield Park, Quebec
  - Lachine, Quebec
  - Laval, Quebec
  - Montreal, Quebec
  - Saint Georges-de-beauce, Quebec
  - Saint-Charles-Borromée, Quebec
  - Saint-Jérôme, Quebec
  - Saint-Lambert, Quebec
  - Ste. Foy, Quebec
  - Sudbury, Quebec
  - Trois-Rivières, Quebec
  - Val-d'Or, Quebec
  - Saskatoon, Saskatchewan
- Germany (10):
  - Aachen
  - Berlin
  - Darmstadt
  - Essen
  - Hamburg
  - Heidelberg
  - Leipzig
  - München
  - Regensburg
  - Ulm
- Poland (7):
  - Elblag
  - Gdansk
  - Krakow
  - Lublin
  - Poznan
  - Warsaw
  - Wroclaw
- Switzerland (3):
  - Geneva
  - Kreuzlingen
  - Zurich

REFERENCES:
- [Derived] Tardif JC, Rhainds D, Brodeur M, Feroz Zada Y, Fouodjio R, Provost S, Boule M, Alem S, Gregoire JC, L'Allier PL, Ibrahim R, Guertin MC, Mongrain I, Olsson AG, Schwartz GG, Rheaume E, Dube MP. Genotype-Dependent Effects of Dalcetrapib on Cholesterol Efflux and Inflammation: Concordance With Clinical Outcomes. Circ Cardiovasc Genet. 2016 Aug;9(4):340-8. doi: 10.1161/CIRCGENETICS.116.001405. Epub 2016 Jul 14. PMID 27418594
- [Derived] Tardif JC, Rheaume E, Lemieux Perreault LP, Gregoire JC, Feroz Zada Y, Asselin G, Provost S, Barhdadi A, Rhainds D, L'Allier PL, Ibrahim R, Upmanyu R, Niesor EJ, Benghozi R, Suchankova G, Laghrissi-Thode F, Guertin MC, Olsson AG, Mongrain I, Schwartz GG, Dube MP. Pharmacogenomic determinants of the cardiovascular effects of dalcetrapib. Circ Cardiovasc Genet. 2015 Apr;8(2):372-82. doi: 10.1161/CIRCGENETICS.114.000663. Epub 2015 Jan 11. PMID 25583994

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dalcetrapib | Placebo
Started | 474 | 462
Completed | 464 | 444
Not Completed | 10 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dalcetrapib | Placebo | Total
Number analyzed (Participants) | 474 | 462 | 936
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.5 (8.48) | 60.4 (8.86) | 60.5 (8.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 127 | 108 | 235
  Male | 347 | 354 | 701

OUTCOME MEASURES:

1. Primary Outcome: Nominal Change From Baseline to Study End in Coronary Percent Atheroma Volume (PAV) of the Target Coronary Artery Assessed by IVUS.
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: Percent Change Atheroma Volume
Arm/Group | Dalcetrapib | Placebo
Number analyzed (Participants) | 474 | 462
Percent Change Atheroma Volume | 0.6 (3.69) | 0.5 (2.01)

2. Primary Outcome: Rate of Change From Baseline to Study End in Carotid Intima-media Thickness (CIMT) Using B-mode Ultrasound
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: mm/year
Arm/Group | Dalcetrapib | Placebo
Number analyzed (Participants) | 363 | 356
mm/year | 0.003 (0.0588) | 0.003 (0.0568)

3. Secondary Outcome: Nominal Changes From Baseline in Minimal Lumen Diameter as Assessed by Quantitative Coronary Angiography
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Dalcetrapib | Placebo
Number analyzed (Participants) | 474 | 462
mm | -0.1 (0.18) | 0.0 (0.10)

4. Secondary Outcome: Blood Lipids, Lipoproteins
Time Frame: Throughout study, 24 months
Population: Data not collected
Arm/Group | Dalcetrapib | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Nominal Changes in Percent Diameter Stenosis as Assessed by Quantitative Coronary Angiography
Time Frame: Throughout Study, 24 months
Measure: Mean (Standard Deviation); unit: Percent Diameter Stenosis
Arm/Group | Dalcetrapib | Placebo
Number analyzed (Participants) | 474 | 462
Percent Diameter Stenosis | 9.2 (20.65) | 4.3 (14.36)

ADVERSE EVENTS:
Arm/Group | Dalcetrapib | Placebo
Serious Adverse Events (participants affected / at risk) | 61/474 | 63/462
Other Adverse Events (participants affected / at risk) | 255/474 | 199/462
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dalcetrapib (N=474) | Placebo (N=462)
Angina Pectoris (Cardiac disorders) | 5 | 3
Angina Unstable (Cardiac disorders) | 2 | 3
Atrial Fibrillation (Cardiac disorders) | 3 | 1
Cardiac Failure Congestive (Cardiac disorders) | 1 | 1
Prinzmetal Angina (Cardiac disorders) | 0 | 2
Sick Sinus Syndrome (Cardiac disorders) | 1 | 1
Atrial Flutter (Cardiac disorders) | 0 | 1
Atrioventricular Block Complete (Cardiac disorders) | 0 | 1
Atrioventricular Block Second Degree (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Sinus Bradycardia (Cardiac disorders) | 1 | 0
Ventricular Extrasystoles (Cardiac disorders) | 0 | 1
Ventricular Tachicardia (Cardiac disorders) | 0 | 1
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Adenolymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Benign Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Brain Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast Cancr Male (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Diffuse Large B-Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant Melonoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant Neoplasm of Ampulla of Vater (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Small Cell Lung Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Thyroid Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Chest Pain (General disorders) | 3 | 7
Non-Cardiac Chest Pain (General disorders) | 1 | 2
Chest Discomfort (General disorders) | 2 | 0
Device Failure (General disorders) | 0 | 1
Medical Device Complication (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Aortic Aneurism (Vascular disorders) | 1 | 1
Hypertension (Vascular disorders) | 1 | 1
Hypertensive Crisis (Vascular disorders) | 1 | 1
Intermittent Claudication (Vascular disorders) | 2 | 0
Arterial Thrombosis Limb (Vascular disorders) | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 1
Hematoma (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
Pneumonia (Infections and infestations) | 3 | 2
Clostridial Infection (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 0 | 1
Wound Infection (Infections and infestations) | 0 | 1
Chronic Obstructive Coronary Disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sleep Apnea Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint Effusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Myositis Ossificans (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 3
Abdominal Pain (Gastrointestinal disorders) | 0 | 1
Crohn's Disease (Gastrointestinal disorders) | 1 | 0
Diarrhea Hemorrhagic (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Hiatus Hernia (Gastrointestinal disorders) | 1 | 0
Rectal Hemorrhage (Gastrointestinal disorders) | 1 | 0
Arterial Injury (Injury, poisoning and procedural complications) | 0 | 1
Foot Fracture (Injury, poisoning and procedural complications) | 1 | 0
Joint Dislocation (Injury, poisoning and procedural complications) | 0 | 1
Limb Traumatic Amputaton (Injury, poisoning and procedural complications) | 0 | 1
Post Procedural Hemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Post Procedural Pulmonary Embolism (Injury, poisoning and procedural complications) | 1 | 0
Wrist Fracture (Injury, poisoning and procedural complications) | 1 | 0
Bile Duct Stone (Hepatobiliary disorders) | 0 | 2
Cholangitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis Acute (Hepatobiliary disorders) | 0 | 1
Hepatic Cirrhosis (Hepatobiliary disorders) | 0 | 1
Carotid Artery Stenosis (Nervous system disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 1 | 0
Monoplegia (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0
Polyneuropathy (Nervous system disorders) | 1 | 0
Calculus Bladder (Renal and urinary disorders) | 0 | 1
Calculus Urinary (Renal and urinary disorders) | 0 | 1
Hematuria (Renal and urinary disorders) | 1 | 0
Renal Colic (Renal and urinary disorders) | 0 | 1
Arteriogram Coronary (Investigations) | 1 | 0
Heart Rate Irregular (Investigations) | 0 | 1
Hepatic Enzyme Increased (Investigations) | 0 | 1
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 2 | 0
Completed Suicide (Psychiatric disorders) | 1 | 0
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Idiopathic Thrombocytopenia Purpura (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Drug Eruption (Skin and subcutaneous tissue disorders) | 1 | 0
Cataract Operation (Surgical and medical procedures) | 1 | 0
Gastrectomy (Surgical and medical procedures) | 1 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dalcetrapib (N=474) | Placebo (N=462)
Diarrhea (Gastrointestinal disorders) | 41 | 27
Back Pain (Musculoskeletal and connective tissue disorders) | 20 | 24
Nasopharyngitis (Infections and infestations) | 27 | 22
Chest Pain (General disorders) | 48 | 36
Headache (Nervous system disorders) | 27 | 23
Dizziness (Nervous system disorders) | 24 | 22
Hypertension (Vascular disorders) | 38 | 19
Angina Pectoris (Cardiac disorders) | 30 | 26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No